CLINICAL TRIAL: NCT04987476
Title: Hétérogénéité Des Tumeurs Rhabdoides : Approches en " Cellules Uniques " Pour Identifier Des Cibles thérapeutiques
Brief Title: Rhabdoid Tumors Cellular Architecture by Single-cell Analyses (InnovRT-2)
Acronym: InnovRT-2
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Curie (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200122; 2021-A00795-36 (Other: ID-RCB Number)
Record Dates: First submitted 2021-07-31; First posted 2021-08-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: ATRT
Keywords: ATRT; SMARCB1; single-cell RNAseq

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ATRT: Children affected by an ATRT at time of surgical resection
  Interventions: Biological: analyzes in singles cells

INTERVENTIONS:
Biological: analyzes in singles cells — genome expression analyzes in single cells

SUMMARY:
The aim is to describe at the cellular level the heterogeneity of rhabdoid tumors, and identify how this diversity influences resistance to treatment.

DETAILED DESCRIPTION:
Rhabdoid tumors are aggressive cancers of infancy. Although frequently chemosensitive at the very beginning, they very often show resistance, suggesting some intra-tumor diversity or plasticity. Moreover, morphological analysis of rhadoid tumors often reveal some variety in tumor cell shapes and immunohistochemical profiling. Altogether, this suggests some intra-tumor heterogeneity, that has been scarcely studied so far.

This project aims to describe the intra-tumor heterogeneity by single-cell sequencing approaches.

After surgical resection, fresh tumor samples will be dissected and analysed using the 10X Chromium technology. Briefly, cells will be grouped in clusters according to their gene expression signalling, and each cluster will be defined in comparison with all other ones. Differential analyses will allow identifying the main characteristic of each cell sub-population. Potential filiations between clusters will be analysed using classical algorithms. The study will be performed on 10 to 15 tumor samples.

ELIGIBILITY:
Inclusion Criteria:

* Aged 0-17 years old
* having a rhabdoid tumor according to clinical and radiological features Or likely having a rhabdoid tumor according to clinical and radiological features
* surgical resection in standard care
* sufficient material for both diagnosis and experimental procedures
* parents' agreement

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children having or likely having a rhabdoid tumor according to clinical and radiological features
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Intra-tumor heterogeneity | Inclusion
  Identification of cell clusters - mean expression (RPKM unit) of gene set signtaures in each bioinformatically defined cluster

SECONDARY OUTCOMES:
Cell clusters recurrent from one sample to the other | Inclusion
  Fraction/percentage of cell clusters defined by primary outcome that are specific to each tumor and those that are shared by several or all samples
Naming of potential targetable gene | Inclusion
  Mean expression (RPKM unit) of targetable genes (defined by the existence of adequate pharmacological inhibitor) in each tumor sample and clusters
Identification of cytotoxic cells | Inclusion
  Conducting therapeutic biological functional tests

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Beccaria, MD, PhD, Pr, Study Director — APHP Assistance Publique des Hôpitaux de Paris
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: No